CLINICAL TRIAL: NCT06426095
Title: Exploring Pedagogical Approaches: A Comparative Analysis of the Efficacy of Instructional Videos and Live Demonstrations in Crown Preparation Training for Preclinical Dental Students
Brief Title: A Comparative Analysis of the Efficacy of Instructional Videos and Live Demonstrations in Crown Preparation Training for Preclinical Dental Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Altamash Institute of Dental Medicine (Other)
Responsible Party: Principal Investigator, Dr Maria Shakoor, Associate Professor, Altamash Institute of Dental Medicine
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: AIDM/ERC/01/2023/02
Record Dates: First submitted 2024-05-08; First posted 2024-05-23 (Actual); Last update posted 2024-05-23 (Actual); Status verified 2024-05

CONDITIONS: Medical Education; Dental; Dental Crown Preparation; Instructional Methods; Training Effectiveness
Keywords: Medical Education; Instruction video; Live Demonstrations

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- instructional video (Experimental): Participants in Group A received access to a specially prepared pre-recorded instructional video detailing the step-by-step process of porcelain-fused-to-metal tooth preparation for molars
  Interventions: Behavioral: Group A (instructional video),
- live demonstrations (Experimental): live demonstrations of the same procedure conducted by the same experienced Prosthodontist to ensure consistency in teaching quality and technique.
  Interventions: Behavioral: Group B (live demonstration)
- hybrid (Experimental): both video and live demonstrations will be given
  Interventions: Behavioral: Group C (hybrid)

INTERVENTIONS:
Behavioral: Group A (instructional video), — Participants in Group A received access to a specially prepared pre-recorded instructional video detailing the step-by-step process of porcelain-fused-to-metal tooth preparation for molars.
  Arms: instructional video
Behavioral: Group B (live demonstration) — Participants in Group B were provided with live demonstrations of the same procedure conducted by the same experienced Prosthodontist to ensure consistency in teaching quality and technique
  Arms: live demonstrations
Behavioral: Group C (hybrid) — Group C received a dual approach, combining instructional video guidance with live demonstrations.
  Arms: hybrid

SUMMARY:
finding the optimal balance between traditional live demonstrations and instructional videos remains a subject of ongoing discussion in dental education. Moreover, integrating a hybrid model that combines the strengths of both methods may offer a comprehensive approach to crown preparation training.

Therefore, this study aims to address this ongoing discussion by investigating the relative effectiveness of traditional live demonstrations, instructional videos, and a hybrid model that merges both approaches. Through an evaluation of dental students' satisfaction and performance with video tutorials and hands-on demonstrations, this research endeavors to shed light on how different instructional methods influence knowledge acquisition within the practical environment.

DETAILED DESCRIPTION:
A randomized controlled single-blind trial was conducted at the Department of Prosthodontics, Altamash Institute of Dental Medicine for a duration of 12 months from 12th Jan' 2023 till 11th Jan' 2024.

Prior approval was obtained from the Ethical Review Committee of Altamash Institute of Dental Medicine (AIDM/ERC/01/2023/02). written consent was obtained from all participants, A simple random sampling technique was used for the recruitment of participants. .

a total of ninety-six final-year BDS students were enrolled in the study. Before allocation, all participants attended a comprehensive lecture on crown preparation principles delivered via a PowerPoint presentation. Following the lecture, participants were randomly assigned to one of three groups: Group A (instructional video), Group B (live demonstrations), or Group C (hybrid)

Participants in Group A will view an instructional video, group B will attend live demonstrations.

Participants in Group C received a dual approach, combining instructional video guidance with live demonstrations.

Before the intervention, all participants across the three groups underwent a pretest consisting of five questions. These questions were designed to gauge participants' readiness and perceptions regarding crown preparation training. Responses were recorded using a Likert scale ranging from 1 to 5, where 1 represented "strongly disagree" and 5 represented "strongly agree".

Following the lecture and demonstrations, participants were provided with an assessment questionnaire comprising six questions aimed at evaluating their comprehension and knowledge regarding porcelain-fused-to-metal tooth preparation.

ELIGIBILITY:
Inclusion Criteria:

* Fourth-year students of Bachelor of Surgery who voluntarily agreed to participate were included in the study.

Exclusion Criteria:

* Exclusion criteria include students who do not provide consent, those absent from tutorials, individuals with prior experience in crown preparation, or students with medical conditions affecting participation.

Ages: 24 Years to 26 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 96 (Actual)
Dates: Start 2023-01-12 (Actual); Primary Completion 2024-01-11 (Actual); Study Completion 2024-01-11 (Actual)

PRIMARY OUTCOMES:
Proficiency in Crown Preparation after instructional Videos and Live Demonstrations i | 12 months
  Proficiency in Crown Preparation: Assessed by a standardized scoring chart evaluating key areas such as preparation axis, axial reduction, anatomic reduction, occlusal convergence, occlusal reduction depth, morphology, quality of axial/occlusal line angles, finish line location, form, continuity, and surface texture. Each area is scored to give a total proficiency score out of 20. Measurements will be taken immediately following the intervention period."
students perception about the demonstration techniques of the three groups | 12 months
  Before the intervention, all participants across the three groups underwent a pretest consisting of five questions. These questions were designed to gauge participants' readiness and perceptions regarding crown preparation training. Specifically, the questions addressed stress levels during preparation, the duration of preclinical training, the effectiveness of lectures and training, and readiness for clinical practice. Responses were recorded using a Likert scale ranging from 1 to 5, where 1 represented "strongly disagree" and 5 represented "strongly agree".

CONTACTS AND LOCATIONS:
Locations (1):
- Altamash Institute of dental medicine, Karachi, Pakistan

REFERENCES:
- [Derived] Abbasi MS, Anis A, Billoo S, Altamash S, Ehsan AA, Omer SA, Ilhan D, Khan Z, Ahmed N, Das G, Mosaddad SA. Exploring pedagogical approaches in crown preparation: a randomized controlled trial comparing the efficacy of instructional videos and live demonstrations. BMC Med Educ. 2025 Apr 3;25(1):480. doi: 10.1186/s12909-025-07060-7. PMID 40181303